CLINICAL TRIAL: NCT01008852
Title: Randomized, Parallel, Double-Blind, Placebo-Controlled Trial To Evaluate The Efficacy And Safety Of SBI-087 In Seropositive Subjects With Active Rheumatoid Arthritis On A Stable Background Of Methotrexate
Brief Title: Study Evaluating The Efficacy And Safety Of SBI-087 In Seropositive Subjects With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Emergent Product Development Seattle LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3227K1-2000; B2261003
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Active Rheumatoid Arthritis
Keywords: rheumatoid arthritis; seropositive; methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — SBI-087

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Treatment Group 1 (Experimental)
  Interventions: Drug: SBI-087
- Treatment Group 2 (Experimental)
  Interventions: Drug: SBI-087
- Treatment Group 3 (Experimental)
  Interventions: Drug: SBI-087
- Treatment Group 4 (Experimental)
  Interventions: Drug: SBI-087
- Treatment Group 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SBI-087 — 200 mg SC Day 1, Placebo Day 15, Placebo Day 84 + Methotrexate
  Arms: Treatment Group 1
Drug: SBI-087 — 200 mg SC Day 1, 200 mg SC Day 15, Placebo Day 84 + Methotrexate
  Arms: Treatment Group 2
Drug: SBI-087 — 200 mg SC Day 1, Placebo Day 15, 200 mg SC Day 84 + Methotrexate
  Arms: Treatment Group 3
Drug: SBI-087 — 200 mg SC Day 1, 200 mg SC Day 15, 200 mg SC Day 84 + Methotrexate
  Arms: Treatment Group 4
Drug: Placebo — Placebo Day 1, Placebo Day 15, Placebo Day 84 + Methotrexate
  Arms: Treatment Group 5

SUMMARY:
This study is designed to evaluate the safety and efficacy of a dose and dosage regimen of SBI-087 in seropositive patients with active Rheumatoid Arthritis, who are on a stable dose of methotrexate.

ELIGIBILITY:
Inclusion Criteria:

* Meets the American College of Rheumatology (ACR) 1987 revised criteria for classification of Rheumatoid Arthritis (RA) for at least 6 months prior to screening
* Active RA as defined by >= 5 swollen and >= 5 tender joints (28-joint count) and at least 1 of the following: C-reactive protein >= 10 mg/L or Erythrocyte Sedimentation Rate >= 28 mm/h
* Must be seropositive as defined by a documented history of rheumatoid factor (RF) or anti-cyclic citrullinated peptide (anti-CCP) positivity
* Must be receiving a stable route and dose of methotrexate (up to 25 mg weekly)

Exclusion Criteria:

* Any significant health problem other than rheumatoid arthritis
* Any clinically significant laboratory abnormalities
* Any prior use of B cell-depleting therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2009-12; Primary Completion 2011-09 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Response as measured by American College of Rheumatology criteria (ACR 20 response) | 16 weeks

SECONDARY OUTCOMES:
ACR Responses, 28 Joint Assessment, Pain Visual Analog Scale (VAS), General Health VAS, Physician and Patient Global Assessments, Morning Stiffness Duration, FACIT-Fatigue, SF-36, HAQ-DI, Hybrid Measure of ACR, ACR-N, DAS-28 and EULAR response | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- United States (20):
  - Pfizer Investigational Site, Paradise Valley, Arizona
  - Pfizer Investigational Site, Palm Desert, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Westlake Village, California
  - Pfizer Investigational Site, Newark, Delaware
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Palm Harbor, Florida
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, Worcester, Massachusetts
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Minot, North Dakota
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Tulsa, Oklahoma
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Jackson, Tennessee
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Clarksburg, West Virginia
- Argentina (2):
  - Pfizer Investigational Site, Buenos Aires, C.a.b.a.
  - Pfizer Investigational Site, C.a.b.a
- Canada (3):
  - Pfizer Investigational Site, Winnipeg, Manitoba
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Pointe-Claire, Quebec
- Pfizer Investigational Site, Providencia, Santiago Metropolitan, Chile
- Hungary (4):
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Gyula
  - Pfizer Investigational Site, Miskolc
  - Pfizer Investigational Site, Szolnok
- Japan (10):
  - Pfizer Investigational Site, Aichi
  - Pfizer Investigational Site, Fukui
  - Pfizer Investigational Site, Fukuoka
  - Pfizer Investigational Site, Hokkaido
  - Pfizer Investigational Site, Hyōgo
  - Pfizer Investigational Site, Kanagawa
  - Pfizer Investigational Site, Miyagi
  - Pfizer Investigational Site, Saitama
  - Pfizer Investigational Site, Shizuoka
  - Pfizer Investigational Site, Tokyo
- Pfizer Investigational Site, Coahulia, Torreon, Mexico
- Poland (5):
  - Pfizer Investigational Site, Warsaw, Poland
  - Pfizer Investigational Site, Działdowo
  - Pfizer Investigational Site, Elblag
  - Pfizer Investigational Site, Sopot
  - Pfizer Investigational Site, Warsaw
- Serbia (3):
  - Pfizer Investigational Site, Belgrade
  - Pfizer Investigational Site, Niška Banja
  - Pfizer Investigational Site, Novi Sad
- Spain (3):
  - Pfizer Investigational Site, A Coruña, A Coruña
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Seville, Sevilla

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3227K1-2000&StudyName=Study%20Evaluating%20The%20Efficacy%20And%20Safety%20Of%20SBI-087%20In%20Seropositive%20Subjects%20With%20Active%20Rheumatoid%20Arthritis